CLINICAL TRIAL: NCT05152342
Title: Reducing Stigma Among Individuals With Addiction and Staff in the Criminal Justice System: A Pilot Feasibility Trial
Brief Title: Reducing Stigma Among Individuals With Addiction and Staff in the Criminal Justice System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Kelly E. Moore (Schirr), Assistant Professor, East Tennessee State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0721.5sd
Record Dates: First submitted 2021-11-05; First posted 2021-12-09 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stigma, Social; Behavior
Keywords: stigma reduction; substance use disorder; criminal involvement
MeSH Terms: conditions — Social Stigma; Behavior; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staff intervention (Experimental): Half day virtual training for staff focusing on stigma reduction strategies.
  Interventions: Behavioral: Stigma Awareness Training for Legal System Staff
- Client intervention (Experimental): Three session virtual therapy group for clients focusing on behavioral strategies to cope with stigma.
  Interventions: Behavioral: Acceptance and Commitment Therapy for self-stigma

INTERVENTIONS:
Behavioral: Stigma Awareness Training for Legal System Staff — Multilevel intervention package addressing stigma associated with substance use and criminal involvement for staff and justice-involved clients enrolled in a diversion treatment program.
  Arms: Staff intervention
Behavioral: Acceptance and Commitment Therapy for self-stigma — Multilevel intervention package addressing stigma associated with substance use and criminal involvement for staff and justice-involved clients enrolled in a diversion treatment program.
  Arms: Client intervention

SUMMARY:
Stigma is one of the most pervasive barriers to addiction care in the U.S. criminal justice (CJ) system. However, there have been no stigma reduction interventions developed for this context. This project addresses this gap with a new multi-level stigma intervention, Combatting Stigma to Aid Reentry and Recovery (CSTARR), for justice-involved people with addiction and criminal justice staff. This intervention will be implemented in 6 (mostly rural) counties in TN for clients and staff in the Tennessee Recovery Oriented Compliance Strategy (TN-ROCS) program, which coordinates multiple CJ sectors (i.e., courts, corrections, probation, treatment) to divert and treat people with addiction. This project aims to 1) examine the feasibility, acceptability, and implementation considerations of integrating CSTARR in the TN-ROCS program, and 2) determine whether CSTARR impacts individual, staff, and program-level outcomes. We aim to recruit 25 stakeholders, 80 clients, and 75 staff over the course of this 18-month project to participate in our intervention and evaluation efforts. Staff and clients will be asked to complete online surveys before and after the intervention, as well as 1- and 3-month follow ups, for which they will receive gift-cards. The overall goal of this project is to examine the feasibility and utility of stigma reduction efforts in the criminal justice system to determine whether they can help facilitate engagement with evidence-based addiction care and improve client and staff outcomes.

DETAILED DESCRIPTION:
Stigma is one of the most pervasive barriers to addiction care in the U.S. criminal justice (CJ) system. Stigmatizing attitudes about addiction, its intersecting conditions (i.e., criminal involvement), and its treatment (i.e., medications for opioid use disorder [MOUD]) are widespread throughout court, corrections, probation, and treatment sectors. These attitudes impact treatment decisions as well as how staff interact with clients. CJ-involved individuals with addiction are aware of this stigma, perceiving negative stereotypes, expecting to be judged, and often feeling ashamed and worthless as a result (i.e., self-stigma). Self-stigma is a robust predictor of treatment avoidance, non-compliance, and dropout in many stigmatized groups, including people with addiction and CJ involvement, making this a critical treatment barrier. Despite the negative consequences of stigma in the CJ system, there are virtually no stigma reduction interventions in this context. Given that the CJ system provides a substantial portion of addiction treatment, and untreated addiction increases risk for relapse, re-arrest, overdose, and other negative outcomes, it is essential to address stigma-related barriers to addiction care.

We drew from existing evidence-based interventions to develop a multi-level stigma intervention, Combatting Stigma to Aid Re-entry and Recovery (CSTARR), that simultaneously targets CJ staff attitudes as well as CJ-involved individuals' ability to cope with stigma in separate client and staff interventions. The staff intervention involves a half-day Stigma Awareness Training, and the client intervention involves a three-session Acceptance and Commitment Therapy for self-stigma group that was adapted to address criminal involvement in addition to addiction stigma. We will deliver both interventions virtually in 6 (primarily rural) Tennessee counties that contain infrastructure called the Tennessee Recovery Oriented Compliance Strategy (TN-ROCS). TN-ROCS coordinates multiple CJ sectors (i.e., courts, corrections, probation, treatment) to divert and treat people with addiction, thus presenting a unique unified system to intervene with stigma at both client and staff levels. Also, select TN-ROCS counties are integrating MOUD services, providing an opportunity to reduce stigma that may ultimately impact MOUD engagement. This project aims to 1) examine the feasibility, acceptability, and implementation considerations of integrating CSTARR in the TN-ROCS program, and 2) determine whether CSTARR impacts individual, staff, and program-level outcomes.

We aim to recruit 25 stakeholders, 80 clients, and 75 staff over the course of this 18-month project to participate in our intervention and evaluation efforts. Staff and clients will be asked to complete online surveys before and after the intervention, as well as 1- and 3-month follow ups, for which they will receive gift-cards. The overall goal of this project is to examine the feasibility and utility of stigma reduction efforts in the criminal justice system to determine whether they can help facilitate engagement with evidence-based addiction care and improve client and staff outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any legal system staff (e.g., judges, attorneys, probation officers, treatment staff, support staff) who work with the Tennessee Recovery Oriented Compliance Strategy (TN-ROCS) program in Sullivan, Jefferson, Grainger, Sevier, Monroe, and McMinn counties are eligible to participate in the staff training.
* Clients who have been accepted into the Tennessee Recovery Oriented Compliance Strategy (TN-ROCS) program in Sullivan, Jefferson, Grainger, Sevier, Monroe, and McMinn counties are eligible to participate in the staff training.

Exclusion Criteria:

* Staff who have not had contact with TN-ROCS clients in the past 90 days are not eligible.
* Clients who are not accepted into the TN-ROCS program, or who become re-incarcerated are not eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Perspectives on Stigma Reduction from Baseline to 3 month follow-up (staff) | Baseline, 1-day, 1-month, 3-months
  24-item internally developed measure that assesses perspectives on stigma and use of stigma reduction strategies among staff, total score ranges from 24 to 216 with higher scores indicating more positive views
Change in Social Distance Scale from Baseline to 3 month follow-up (staff) | Baseline, 1-day, 1-month, 3-months
  5-item adapted measure that assesses desired social distance from people with a criminal and addiction history, total score ranges from 5-25 with higher scores indicating less desired social distance
Change in Difference and Disdain Scale from Baseline to 3 month follow-up (staff) | Baseline, 1-day, 1-month, 3-months
  9-item adapted measure that assesses how staff view people who have substance use problems and criminal involvement, total score ranges from 9-81 with higher scores indicating more differences/disdain
Change in Substance Use Self-Stigma Scale from Baseline to 3 month follow-up (client) | Baseline, 1-day, 1-month, 3-months
  41-item measure that assess how clients view themselves because of their criminal involvement and substance use problems, total score ranges from 41 to 205 with higher scores indicating more self-stigma
Change in Internalized Shame Scale from Baseline to 3 month follow-up (client) | Baseline, 1-day, 1-month, 3-months
  24-item measures that assesses internalized shame, total score ranges from 40-120, with higher scores indicating more internalized shame
Change in Self-efficacy from Baseline to 3 month follow-up (client) | Baseline, 1-day, 1-month, 3-months
  4-item measure that assesses clients' self-efficacy for navigating stigma stressors, total score ranges from 4-40 with higher scores indicating more self-efficacy

SECONDARY OUTCOMES:
Change in Attitudes Toward Prisoners Scale from Baseline to 3 month follow-up (staff) | Baseline, 1-day, 1-month, 3-months
  36-item measure that assesses attitudes, beliefs, and negative stereotypes about people with criminal involvement, total score ranges from 36 to 180 with high scores indicating more stigmatizing attitudes
Change in Dual-Relationship Inventory from Baseline to 3 month follow-up (staff) | Baseline, 1-day, 1-month, 3-months
  9-item measure that assesses how staff view and treat the justice-involved people they oversee, total scores range from 9 to 63 with higher scores indicating better relationships
Change in Treatment Experiences Scale from Baseline to 3 month follow-up (client) from Baseline to 3 month follow-up (client) | Baseline, 1-day, 1-month, 3-months
  13-item adapted measure that assesses how clients feel about their ability to complete treatment, total scores range from 13 to 130 with higher scores indicating more confidence in treatment
Change in Dual-Relationship Inventory from Baseline to 3 month follow-up (client) | Baseline, 1-day, 1-month, 3-months
  9-item adapted measure that assesses how justice-involved clients feel staff view and treat them, total scores range from 9 to 63 with higher scores indicating better relationships

OTHER OUTCOMES:
Implementation outcome (staff) | 1-day
  12-item internally developed measure that assesses how appropriate, useful, and relevant the stigma training is, total scores range from 12 to 60 with higher scores indicating more acceptability
Implementation outcome (client) | 1-day
  12-item internally developed measure that assesses how appropriate, useful, and relevant the stigma group is, total scores range from 12 to 60 with higher scores indicating more acceptability

CONTACTS AND LOCATIONS:
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

REFERENCES:
- [Derived] Moore KE, Johnson JE, Luoma JB, Taxman F, Pack R, Corrigan P, Hart J, Slone JD. A multi-level intervention to reduce the stigma of substance use and criminal involvement: a pilot feasibility trial protocol. Health Justice. 2023 May 15;11(1):24. doi: 10.1186/s40352-023-00224-x. PMID 37184615